CLINICAL TRIAL: NCT01125475
Title: A Scandinavian Non-interventional Study of Adherence to RebiSmart Administered Rebif New Formulation (RNF) Treatment in Relapsing Remitting Multiple Sclerosis (RRMS) Subjects: the ScanSmart Study
Brief Title: A Scandinavian Non-interventional Study of Adherence to RebiSmart Administered Rebif New Formulation (RNF) Treatment in Relapsing Remitting Multiple Sclerosis (RRMS) Subjects
Acronym: SCANSMART
Status: Completed | Type: Observational
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck Serono Norway (Industry); Smerud Medical Research International AS (Other)
Responsible Party: Sponsor
Other Study IDs: EMR 701068-521
Record Dates: First submitted 2010-05-17; First posted 2010-05-18 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2012-09

CONDITIONS: Relapsing Remitting Multiple Sclerosis (RRMS)
Keywords: Relapsing Remitting Multiple Sclerosis; RebiSmart; Rebif; Adherence
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: RebiSmart — Treatment with Rebif New Formulation using RebiSmart.

SUMMARY:
The primary objective is to determine adherence to Rebif® New Formulation administered by RebiSmart during 12 weeks of therapy in patients with RRMS.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between 18 and 65 years of age
* Have relapsing-remitting multiple sclerosis (RRMS) according to the revised McDonald Criteria (2005)
* Having an expanded disability status scale (EDSS) of less than 6 at the screening visit or within 2 months prior to the screening visit
* Stable treatment (defined as treatment after titration period) with RebiSmart administered Rebif new formulation (RNF) 22/44 mcg subcutaneously thrice a week for a minimum of 4 weeks prior to inclusion
* Previously treated with disease modifying drugs (DMDs) for a minimum of 6 months prior to the screening visit
* Female subjects must be neither pregnant nor breast-feeding and must lack child-bearing potential as defined by either:

  * Post-menopausal or surgically sterile; or
  * Using a highly effective method of contraception for the duration of the study. This is defined as a method that results in a low failure rate (i.e. less than 1% per year) when used consistently and correctly , and includes for instance implants, injectables, combined oral contraceptives, intra-uterine device (IUD), sexual abstinence or vasectomized partner
* Have a scheduled visit 12 weeks after the inclusion visit
* Willing and able to comply with the protocol for the duration of the study
* Have given written informed consent

Exclusion Criteria:

* Have had a relapse within 30 days prior to the first visit
* Have any contra-indications to treatment with Interferon-beta 1a according to Summary of Product Characteristics
* Have any other significant disease that in the Investigator's opinion would exclude the subject from the trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Neurology Clinics at Danish and Norwegian hospitals (single treatment group)
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2010-08; Primary Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Adherence assessment | 12 weeks
  Adherence to RNF administered by RebiSmart during 12 weeks of therapy in patients with RRMS

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Serono Norway
Locations (1):
- Sandvika Nevrosenter, Sandvika, Sandviksveien 178, Norway